CLINICAL TRIAL: NCT03202316
Title: A Phase II Study of Triple Combination of Atezolizumab + Cobimetinib + Eribulin (ACE) or Atezolizumab + Eribulin (AE) in Patients With Recurrent/Metastatic Inflammatory Breast Cancer
Brief Title: Atezolizumab, Cobimetinib, and Eribulin in Treating Patients With Chemotherapy Resistant Metastatic Inflammatory Breast Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-0890; NCI-2017-01601 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2016-0890 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2017-06-27; First posted 2017-06-28 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Recurrent Breast Inflammatory Carcinoma; Stage IV Breast Inflammatory Carcinoma
MeSH Terms: conditions — Inflammatory Breast Neoplasms | interventions — atezolizumab; cobimetinib; eribulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort I (atezolizumab, cobimetinib, eribulin) (Experimental): Patients receive atezolizumab IV over about 30-60 minutes every 2 weeks, cobimetinib PO daily for 3 weeks on, 1 week off for 4 weeks of the safety lead-in course. Patients then receive atezolizumab IV over about 30-60 minutes every 2 weeks, cobimetinib PO daily for 3 weeks on, 1 week off, and eribulin IV over 2-5 minutes on days 1 and 8 of cycles 1-4. Cycles 1-4 repeat every 21 days and subsequent cycles with atezolizumab and cobimetinib repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Atezolizumab; Drug: Cobimetinib; Drug: Eribulin; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study
- Cohort II (atezolizumab, eribulin) (Experimental): Patients receive atezolizumab IV over about 30-60 minutes every 3 weeks for cycles 1-6 and every 4 weeks for subsequent cycles, and eribulin IV over 2-5 minutes on days 1 and 8 of cycles 1-6. Cycles 1-6 repeat every 21 days and subsequent cycles with atezolizumab repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Atezolizumab; Drug: Eribulin; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study

INTERVENTIONS:
Drug: Atezolizumab — Given IV
  Other Names: MPDL 3280A; MPDL 328OA; MPDL-3280A; MPDL3280A; MPDL328OA; RG7446; RO5541267; Tecentriq
Drug: Cobimetinib — Given PO
  Other Names: Cotellic; GDC-0973; MEK Inhibitor GDC-0973; XL518
  Arms: Cohort I (atezolizumab, cobimetinib, eribulin)
Drug: Eribulin — Given IV
  Other Names: ER-086526
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase II trial studies how well atezolizumab, cobimetinib, and eribulin work in treating patients with inflammatory breast cancer that has spread to other places in the body (metastatic). Immunotherapy with monoclonal antibodies, such as atezolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Cobimetinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as eribulin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving atezolizumab, cobimetinib, and eribulin may work better in treating patients with inflammatory breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine ORR (overall response rate) of metastatic inflammatory breast cancer (BC) (mIBC) patients treated with this proposed combinatorial atezolizumab, cobimetinib, and eribulin (ACE) therapy via phase II. (ACE, Cohort I) II. To determine ORR (overall response rate) for double combination of atezolizumab and eribulin (AE). (AE, cohort II)

SECONDARY OBJECTIVES:

I. To further characterize the safety and tolerability of atezolizumab + cobimetinib + eribulin.

II. To further characterize the safety and tolerability of atezolizumab + eribulin.

III. To determine CBR (clinical benefit rate): (stable disease [SD] + complete response [CR] + partial response [PR] >= 24 weeks).

III. To determine the duration of response (DOR). IV. To determine progression free survival (PFS). V. To determine 2 years overall survival (OS).

EXPLORATORY OBJECTIVES:

I. To determine the progressive disease (PD) biomarker changes induced by combinatorial therapy using liquid and tissue based assays to investigate microenvironment via multiplex imaging, proportional study of T cells: CD3, CD8 composition and change, macrophage (M1 and M2), PD-L1 expression on circulating tumor cell (CTC).

II. To determine the immune pathway related biomarker changes induced by combinatorial therapy via multiplex serum cytokine assays.

III. This translational biomarker assays will be done based on collaboration with plasma based ribonucleic acid (RNA) sequencing (RNA-seq) in collaboration with Lambowitz laboratory (lab) (University of Texas at Austin [UT Austin]), Oncomine next-generation sequencing (NGS) study on tumor/circulating tumor deoxyribonucleic acid (ctDNA) with Wistuba lab, and bioinformatics with Futreal lab.

OUTLINE:

COHORT I: Patients receive atezolizumab intravenously (IV) over about 30-60 minutes every 2 weeks, cobimetinib orally (PO) daily for 3 weeks on, 1 week off for 4 weeks of the safety lead-in course. Patients then receive atezolizumab IV over about 30-60 minutes every 2 weeks, cobimetinib PO daily for 3 weeks on, 1 week off, and eribulin IV over 2-5 minutes on days 1 and 8 of cycles 1-4. Cycles 1-4 repeat every 21 days and subsequent cycles with atezolizumab and cobimetinib repeat every 28 days in the absence of disease progression or unacceptable toxicity.

COHORT II: Patients receive atezolizumab IV over about 30-60 minutes every 3 weeks for cycles 1-6 and every 4 weeks for subsequent cycles, and eribulin IV over 2-5 minutes on days 1 and 8 of cycles 1-6. Cycles 1-6 repeat every 21 days and subsequent cycles with atezolizumab repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of the study treatment, patients are followed for 3 months and then every 6 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form (ICF) and comply with the requirements of the study protocol
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Confirmed diagnosis of inflammatory breast cancer according to international consensus criteria: (1) onset: rapid onset of breast erythema, edema, and/or peau d'orange, and/or warm breast, with or without an underlying breast mass (2) duration: history of such findings no more than 6 months (3) extent: erythema occupying at least 1/3 of whole breast (4) pathology: pathologic confirmation of invasive carcinoma
* Patients with recurrent or metastatic IBC after standard systemic therapy are eligible; patients who have disease progression while receiving standard anthracycline or taxane based neoadjuvant therapy are also eligible. a. patients with HER2-positive disease must have had at least 2 lines of anti-HER2 therapy, including Perjeta and Kadcyla; b. prior eribulin treatment is allowed
* At least one metastatic lesion amendable for biopsy (core, punch, or fine needle aspiration [FNA]); if the patient only has lymph nodes, these are considered amenable but will not be biopsied
* At least one site of measurable disease (per Response Evaluation Criteria in Solid Tumors [RECIST] 1.1), local or distant
* Any estrogen receptor (ER), progesterone receptor (PR), HER2 status
* Absolute neutrophil count (ANC) >= 1500 cells/uL (obtained within 14 days prior to the first study treatment [PD window day 1])
* White blood cell (WBC) counts > 2500/uL (obtained within 14 days prior to the first study treatment [PD window, day 1])
* Lymphocyte count >= 300/uL (obtained within 14 days prior to the first study treatment [PD window day 1])
* Platelet count >= 100,000/uL (obtained within 14 days prior to the first study treatment [PD window day 1])
* Hemoglobin >= 9.0 g/dL (obtained within 14 days prior to the first study treatment [PD window day 1])
* Total bilirubin =< 1.5 x upper limit of normal (ULN) with the following the exception: Patients with known Gilbert disease who have serum bilirubin level =< 3 x ULN may be enrolled (obtained within 14 days prior to the first study treatment [PD window, day 1])
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x ULN with the exception: Patients with liver involvement: AST and/or ALT =< 5 x ULN (obtained within 14 days prior to the first study treatment [PD window, day 1])
* Alkaline phosphatase =< 2.5 x ULN with the exception: Patients with documented liver involvement or bone metastases: alkaline phosphatase =< 5 x ULN (obtained within 14 days prior to the first study treatment [PD window, day 1])
* Serum creatinine =< 1.5 x ULN or creatinine clearance >= 50 mL/min on the basis of the Cockcroft-Gault glomerular filtration rate estimation (obtained within 14 days prior to the first study treatment [PD window, day 1])
* For women of childbearing potential or male subjects: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods that result in a failure rate of < 1% per year, during the treatment period and for at least 5 months after the last dose of treatment
* International normalized ratio (INR) and activated partial thromboplastin time (aPTT) =< 1.5 x ULN for patients who do not receive therapeutic anticoagulation
* Patients receiving therapeutic anticoagulation (such as low-molecular-weight heparin or warfarin) should be on a stable dose
* Left ventricular ejection fraction >= 50% measured by multigated acquisition (MUGA) scan or echocardiogram

Exclusion Criteria:

* Any approved anticancer therapy for treatment purpose is not allowed, or need to be stopped at least 2 weeks prior to initiation of study treatment; however, the following are allowed: a. endocrine therapy (selective estrogen receptor modulator [SERM], aromatase inhibitor, fulvestrant) b. palliative radiotherapy for bone metastases > 1 week prior to study treatment c. stable brain metastasis and asymptomatic treated central nervous system (CNS) metastases are allowed, patient must show stable disease by CNS radiographic study >= 4 weeks from completion of radiotherapy and >= 2 weeks from discontinuation of corticosteroids
* Adverse events (AEs) from prior anticancer therapy that have not resolved to grade =< 1 except for alopecia and neuropathy
* Grade 3 or above neuropathy induced from prior treatment, that is not resolved to grade 2 or below despite best supportive care
* Known clinically significant liver disease, including active viral, alcoholic, or other hepatitis; cirrhosis; fatty liver; and inherited liver disease
* Pregnancy, lactation, or breastfeeding
* Known hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies
* Inability to comply with study and follow-up procedures
* Active or history of autoimmune disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjogren's syndrome, Guillain-Barre syndrome, or multiple sclerosis, with the following exception: a. patients with a history of autoimmune hypothyroidism who are on thyroid replacement hormone are eligible for the study; b. patients with controlled type 1 diabetes mellitus who are on an insulin regimen are eligible for the study; c. patients with eczema, psoriasis, lichen simplex chronicus of vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis would be excluded) are permitted provided that they meet the following conditions are met: i. rash must cover < 10% of body surface area.; ii. disease is well controlled at baseline and requires only low-potency topical corticosteroids; iii. no occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high potency or oral corticosteroids within the previous 12 months
* Acute exacerbations of underlying condition within the last 12 months (requiring psoralen plus ultraviolet A radiation [PUVA], methotrexate, retinoids, biologic agents, oral calcineurin inhibitors; high potency or oral steroids)
* Known history of idiopathic pulmonary fibrosis, pneumonitis (including drug induced), organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia, etc.), or evidence of active pneumonitis on screening chest computed tomography (CT) scan:

  * History of radiation pneumonitis in the radiation field (fibrosis) is permitted
* Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk from treatment complications
* Known history of human immunodeficiency virus (HIV) infection or active hepatitis B (chronic or acute) or hepatitis C infection; but: a. patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction (PCR) is negative for hepatitis C virus (HCV) RNA; b. patients with past or resolved hepatitis B infection (defined as having a negative hepatitis B surface antigen [HBsAg] test and a positive anti-HBc [antibody to hepatitis B core antigen] antibody test) are eligible, but should sample for hepatitis B virus (HBV) DNA and referral to virologist to monitor for HBV reactivation
* Active tuberculosis based on history, symptoms, physical exam, imaging
* Severe infections within 4 weeks prior to study treatment, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia
* Signs or symptoms of infection within 2 weeks prior to study treatment
* Received oral or IV antibiotics within 2 weeks prior to study treatment

  * Patients receiving prophylactic antibiotics (e.g., for prevention of a urinary tract infection or chronic obstructive pulmonary disease) are eligible
* Major surgical procedure within 28 days prior to study treatment or anticipation of need for a major surgical procedure during the course of the study
* Patients must agree not to receive any live, attenuated influenza vaccine (e.g., FluMist) within 28 days prior to receiving study treatment, during treatment or within 5 months following the last dose of atezolizumab
* Malignancies other than the disease under study within 5 years prior to study treatment, with the exception of those with a negligible risk of metastasis or death and with expected curative outcome (such as adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, or ductal carcinoma in situ treated surgically with curative intent) or undergoing active surveillance per standard-of-care management (e.g., chronic lymphocytic leukemia Rai Stage 0)
* COBIMETINIB-SPECIFIC EXCLUSION CRITERIA (ONLY FOR COHORT I):
* History of or evidence of retinal pathology on ophthalmologic examination that is considered a risk factor for neurosensory retinal detachment/central serous chorioretinopathy (CSCR), retinal vein occlusion (RVO), or neovascular macular degeneration
* Patients will be excluded if they currently have the following risk factors for retinal vein occlusion (RVO): (1) uncontrolled glaucoma with intra-ocular pressures >= 21 mmHg (2) serum cholesterol >= grade 2 (3) hypertriglyceridemia >= grade 2 (4) hyperglycemia (fasting) >= grade 2
* Patients with congestive heart failure, congenital long QT syndrome; bradyarrhythmias, drugs known to prolong the QT interval unless the principal investigator and/or attending physician deems the risk for QT prolongation to be low
* The following foods/supplements are prohibited at least 7 days prior to initiation of and during study treatment: (1) St. John's wort or hyperforin (potent CYP3A4 enzyme inducer) (2) grapefruit juice (potent cytochrome P450 CYP3A4 enzyme inhibitor)
* ATEZOLIZUMAB-RELATED EXCLUSION CRITERIA:
* Prior treatment with anti-PD-1, or anti-PD-L1 therapeutic antibody or pathway targeting agents: (a) patients who have received prior treatment with anti·CTLA-4 may be enrolled, provided the following requirements are met: (i) minimum of 12 weeks from the first dose of anti-CTLA-4 and > 6 weeks from the last dose; (ii) no history of severe immune-related adverse effects from anti-CTLA 4 (National Cancer Institute [NCI] Common Terminology for Cancer Adverse Effects CTCAE] grade 3 and 4)
* Treatment with systemic immunostimulatory agents (including but not limited to interferon [IFN]-a or interleukin [IL]-2) within 6 weeks or five half-lives of the drug (whichever is shorter) prior to study treatment
* Treatment with investigational agent within 4 weeks prior to study treatment (or within five half lives of the investigational product, whichever is longer)
* Treatment with systemic immunosuppressive medications (including but not limited to prednisone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [anti-TNF] agents) within 2 weeks prior to study treatment; a. patients who have received acute, low dose, systemic immunosuppressant medications (e.g., a one-time dose of dexamethasone for nausea) may be enrolled; b. the use of inhaled corticosteroids and mineralocorticoids (e.g., fludrocortisone) for patients with orthostatic hypotension or adrenocortical insufficiency is allowed
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
* Patients with prior solid organ transplantation on anti-immunosuppressant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2017-08-11 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | Up to 2 years
  Calculated per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. ORR is defined as the rate of patients who achieved partial response or complete response as the best response. All tumor response will be evaluated by RECIST 1.1. The ORR will be estimated along with 95% confidence intervals. Logistic regression model will be used to assess other variables' effect on the best ORR.

SECONDARY OUTCOMES:
Incidence of dose limiting toxicity (DLT) of cobimetinib and atezolizumab (safety lead-in) | Up to 7 weeks
  Evaluated according to Common Terminology Criteria for Adverse Events version 4.0. DLT is defined as any treatment-emergent adverse events (AEs) occurring during the first 7 weeks (progressive disease window and cycle 1) not clearly attributable to a cause other than the study drugs.
Clinical benefit rate (CBR) | Up to 2 years
  Defined as the rate of patients who achieved complete response, partial response, and stable disease for >= 24 weeks as the best response of treatment. CBR is defined as the rate of patients who achieved complete response, partial response, and stable disease for >= 24 weeks as the best response of treatment.
Duration of response (DOR) | Up to 2 years
  Defined as the period measured from the date of the first occurrence of a complete response (CR) or partial response (PR) (whichever status is recorded first) until the first date that progressive disease or death is documented. Patients who have not progressed and who have not died by the date of data cutoff for analysis will be censored at the time of last tumor assessment date. If no tumor assessments were performed after the date of the first occurrence of a CR or PR, DOR will be censored at the date of the first occurrence of a CR or PR plus remaining stable response from that time point.
Progression free survival (PFS) | From date of treatment start until date of first documented disease progression or death, whichever occurs first, assessed up to 2 years
  Data from patients who have not experienced disease progression or death will be censored at the last tumor assessment date and known to be free of disease progression. Data from patients with no post-baseline tumor assessment will be censored at the treatment start date plus 1 day. PFS will be estimated using the Kaplan-Meier method and the comparison between or among patient's characteristic groups will be evaluated by log-rank test. The Cox regression model may be applied to assess the effect of covariates of interest on PFS.
Overall survival (OS) | At 2 years
  OS will be estimated using the Kaplan-Meier method and the comparison between or among patient's characteristic groups will be evaluated by log-rank test. The Cox regression model may be applied to assess the effect of covariates of interest on OS.
Pharmacodynamic markers | Up to 2 years
  Biomarker changes induced by combinatorial therapy using liquid and tissue based assays to investigate microenvironment via multiplex imaging, proportional study of T cells: CD3, CD8 composition and change, macrophage (M1and M2), PD-L1 expression on circulating tumor cell will be measured. Immune pathway related biomarker changes induced by combinatorial therapy via multiplex serum cytokine assays will be determined. This translational biomarker assays will be done based on collaboration with plasma based ribonucleic acid (RNA) sequencing (RNA-seq) in collaboration with Lambowitz laboratory (lab), Oncomine next-generation sequencing (NGS) study on tumor/circulating tumor deoxyribonucleic acid (ctDNA) with Wistuba lab, and bioinformatics with Futreal lab.
Incidence of adverse events | Up to 2 years
  Detailed safety and tolerability of the combination of cobimetinib, atezolizumab, and eribulin will be assessed. Toxicity data will be summarized by frequency tables.

CONTACTS AND LOCATIONS:
Overall Officials: Vicente Valero, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org